CLINICAL TRIAL: NCT06069388
Title: Benefits of Diaphragm Treatment in Reducing Low Back Pain in Patients With Mechanical Lumbar Pain
Brief Title: Effectiveness of Diaphragm Treatment in Reducing Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Lourdes María Fernández Seguín, Assistant Professor. Physiotherapy Department, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIAFRAGMA
Record Dates: First submitted 2023-09-18; First posted 2023-10-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain, Mechanical
Keywords: low back pain; diaphragm; lumbar pain; physiotherapy; conventional; treatment
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm technique (Experimental): The continuity between the diaphragm and the lumbar spine demonstrates the existence of an anatomical and functional connection between them. Changes in the mobility of the diaphragmatic domes in addition to improvement in spirometric parameters when carrying out a diaphragm stretching technique. This makes us think that the mobility of the lumbar spine may be compromised by diaphragm dysfunction.
  Interventions: Procedure: diaphragm technique; Procedure: conventional therapy
- conventional physiotherapy (Active Comparator): Application of the tetrapolar transcutaneous electrical neurostimulation (TENS) device with the "I-tech Mio-care" equipment in the analgesia program with an intensity of between 10-20 milliamps, according to the patient's tolerance, with an application time of 15 minutes in the lumbar paravertebral area on both sides. 250w infrared lamp at a distance of 1m from the patient, with an application time of 10 minutes. Ultrasound on the quadratus lumborum muscle area with a frequency of 1Mhz, at an intensity of 1.2w/cm2 and with an application time of 10 minutes. Ischemic compression and analytical stretching of the quadratus lumborum, multifidus and iliocostalis muscles, constant pressure with the thumb on each muscular trigger point (MTrP) for between 30 s and 2 min the intensity of the pressure will be adjusted to a level at which each subject reports "comfortable pain", that is, between the pain threshold and the maximum tolerable pain
  Interventions: Procedure: conventional therapy

INTERVENTIONS:
Procedure: diaphragm technique — The patient will be placed in a supine position with knees bent on a cushion. The therapist will position himself oriented from the patient's head towards his feet. The therapist will make contact with the ulnar edge of his hands on the lower edge of the last ribs. It will be pulled cephalad during the inspiratory time, opening the rib cage laterally. Traction will be maintained during expiratory time and repeated during a cycle of 10 breaths.
  Arms: Diaphragm technique
Procedure: conventional therapy — The patient will be placed in a supine position with knees bent on a cushion. The therapist will position himself oriented from the patient's head towards his feet. The therapist will make contact with the ulnar edge of his hands on the lower edge of the last ribs. It will be pulled cephalad during the inspiratory time, opening the rib cage laterally. Traction will be maintained during expiratory time and repeated during a cycle of 10 breaths.

SUMMARY:
Objective: Determine the benefits of including a Stretching technique of the anterior part of the diaphragm in the supine position in the conventional physiotherapy treatment protocol applied to insurance company patients with mechanical low back pain.

design: The aim is to carry out an experimental, analytical, prospective, longitudinal, randomized, single-blind study with a blinded evaluator, with an experimental group (EG) to which a manual technique on the diaphragm will be included in the conventional physiotherapy treatment (manual therapy and electrotherapy). and a control group (CG) to which only conventional physiotherapy treatment is administered.

Subject: Patient diagnosed with subacute or chronic mechanical low back pain by a specialist doctor and who has attended in "Fisioclinic" physiotherapy clinic, Older than 18 years-old, Indistinct sex, Diaphragm dysfunction.

Methods: it is proposed to carry out a study in which two groups of subjects with mechanical low back pain will be compared. One group will receive conventional physiotherapy, with electrotherapy and massage therapy, while the other group will receive the same conventional physiotherapy plus a specific technique aimed at the diaphragm muscle. Ten treatment sessions will be carried out daily from Monday to Friday. Different variables will be evaluated using scientifically validated methods, such as manual diagnostic tests for lumbar mobility, algometry to measure muscle pain, cirtometry to evaluate chest mobility, validated questionnaires for quality of life and spirometry to measure respiratory parameters. These variables will be measured before and after each treatment session and later a week, a month and four months after the last intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with subacute or chronic mechanical low back pain by a specialist doctor and who has attended in "Fisioclinic" physiotherapy clinic.

  * Older than 18 years-old.
  * Indistinct sex.
  * Diaphragm dysfunction.

Exclusion Criteria:

* Any surgical intervention on the upper and lower limbs, head, spine, thorax or abdomen at any time in their lives, with a visible anatomy cause on imaging tests.
* Any pathology of non-mechanical origin, such as inflammatory, infectious, tumorous, neurological, traumatic processes and bone diseases in the lumbar spine.
* Having received analgesic or anti-inflammatory medical treatment for pain in a period of less than two weeks.
* Pregnant women, including the breastfeeding period.
* Patients receiving chemotherapy or radiotherapy.
* Basic systemic disease of rheumatic origin (for example, arthritis, osteoarthritis, gout and psoriasis).
* Implanted electronic devices.
* Drug or alcohol abuse, analgesic or sedative therapy and use of medications that affect the central nervous system (for example, antidepressants, anxiolytics and anticonvulsants).
* Patients who have previous experience with manual treatment of the diaphragm.
* Patients with high work activity.
* Outside the age range for the study.
* Refusal to participate in the study.
* Refusal to complete and sign the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Schober test | baseline, pre-intervention/procedure/surgery
  The Schober test measures the degree of elasticity of the spine, the coxofemoral joints or the hamstring muscles, taking into account that the overall mobility of the spine depends on all the segments that constitute it. It will be performed with the patient standing with his arms along the trunk. The therapist will stand on one side of the patient in a double feint facing towards him. With the help of a marker, the therapist makes a horizontal mark at the level of the S1 vertebra and another 10 cm above this first one. He asks the patient to lean forward and measures the distance between both marks. Next, he asks you again to extend the trunk and measures this distance again.
Fingers-Floor Distance (DDS) test | baseline, pre-intervention/procedure/surgery
  This test is used to assess the elasticity of the spine. It will be performed with the patient standing with feet together and knees fully extended. The therapist will stand next to the patient in a squatting position to be able to make the resulting measurement with the help of a measuring tape. The therapist asks the patient to anteflexion the spine so that his arms, hands and fingers are fully extended and relaxed forward. In the same way, at the end of anteflexion the therapist must measure the distance between the tips of the fingers and the floor with a tape measure. If pain appears in the second part of the movement, one can think of the existence of a dysfunction of the lumbar spine or the sacroiliac joints. Likewise, if the symptoms are accentuated in the third part of anteflexion, the therapist may think of an alteration of the upper lumbar or thoracic spine.
Measurement of thoracic expansion | baseline, pre-intervention/procedure/surgery
  It can be used as a method of evaluating the expansion of diaphragmatic breathing to quantify possible alterations in thoracic capacity and abdominal and chest wall compliance achieved by all expiratory and inspiratory muscles. By recording the expansion of the rib cage with a tape measure over the second intercostal space (axillary level), the xiphoid process, and the midpoint between the xiphoid process and the umbilicus (abdominal level), proficiency in diaphragmatic breathing can be demonstrated.It will be evaluated with cirtometry using a simple measuring tape, marked in centimeters, around the thorax and abdomen. With the patient standing and with their hands on their head, the patient will be asked to "inhale as much as possible" and "exhale as much as possible."
Pressure pain threshold (PPT) of the five lumbar vertebrae, quadratus lumborum and lumbar paravertebral | baseline, pre-intervention/procedure/surgery
  using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer (quantitative v.), in the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L312. In the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L3. PPT measurements will be performed manually gradually until the patient begins to feel pain. This process will be carried out three times in the same place and within an interval of 30 to 60 s, using the average of these three measurements.
Measurement of respiratory parameters through spirometry | baseline, pre-intervention/procedure/surgery
  First the subject is seated, the patient holds the spirometer horizontally in his right hand with the screen pointing upward. He puts the spirometer near his mouth and presses the operation button. You will hear a short beep. At the second beep, the subject takes in as much air as possible. Then place the mouthpiece of the spirometer in your mouth and blow as hard as you can for at least 1.5 seconds. The measurement will be repeated at least three times. One-minute intervals will be applied between these measurements to avoid fatigue of the respiratory muscles in the short term. We will measure the parameters of forced expiratory volume at one second (FEV1) and forced vital capacity (CVF).
Evaluation of quality of life using the SF-12 life questionnaire. (quantitative v.) | baseline, pre-intervention/procedure/surgery
  The health-related quality of life questionnaire Short-Form 12-item (SF-12), which will be applied to determine the measure of health-related quality of life in the direct score and the optimal normalized values to evaluate the domains of physical and mental health. The evaluator will explain each of the items on the scales to the patient, and the patient will complete them in paper format in the presence of the evaluator to resolve any questions they may have. Later the evaluator will extract the scores. Scale of 12 questions in which each item of the scale evaluates different aspects on a scale from 0 (no quality of life) to 100 (highest quality of life). 100 being a result that indicates optimal health and 0 reflecting a state of very bad health.

SECONDARY OUTCOMES:
Schober test | immediately after the intervention/procedure/surgery
  The Schober test measures the degree of elasticity of the spine, the coxofemoral joints or the hamstring muscles, taking into account that the overall mobility of the spine depends on all the segments that constitute it. It will be performed with the patient standing with his arms along the trunk. The therapist will stand on one side of the patient in a double feint facing towards him. With the help of a marker, the therapist makes a horizontal mark at the level of the S1 vertebra and another 10 cm above this first one. He asks the patient to lean forward and measures the distance between both marks. Next, he asks you again to extend the trunk and measures this distance again.
Fingers-Floor Distance (DDS) test | immediately after the intervention/procedure/surgery
  This test is used to assess the elasticity of the spine. It will be performed with the patient standing with feet together and knees fully extended. The therapist will stand next to the patient in a squatting position to be able to make the resulting measurement with the help of a measuring tape. The therapist asks the patient to anteflexion the spine so that his arms, hands and fingers are fully extended and relaxed forward. In the same way, at the end of anteflexion the therapist must measure the distance between the tips of the fingers and the floor with a tape measure. If pain appears in the second part of the movement, one can think of the existence of a dysfunction of the lumbar spine or the sacroiliac joints. Likewise, if the symptoms are accentuated in the third part of anteflexion, the therapist may think of an alteration of the upper lumbar or thoracic spine.
Measurement of thoracic expansion | immediately after the intervention/procedure/surgery
  It can be used as a method of evaluating the expansion of diaphragmatic breathing to quantify possible alterations in thoracic capacity and abdominal and chest wall compliance achieved by all expiratory and inspiratory muscles. By recording the expansion of the rib cage with a tape measure over the second intercostal space (axillary level), the xiphoid process, and the midpoint between the xiphoid process and the umbilicus (abdominal level), proficiency in diaphragmatic breathing can be demonstrated.It will be evaluated with cirtometry using a simple measuring tape, marked in centimeters, around the thorax and abdomen. With the patient standing and with their hands on their head, the patient will be asked to "inhale as much as possible" and "exhale as much as possible."
Pressure pain threshold (PPT) of the five lumbar vertebrae, quadratus lumborum and lumbar paravertebral | immediately after the intervention/procedure/surgery
  using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer (quantitative v.), in the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L312. In the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L3. PPT measurements will be performed manually gradually until the patient begins to feel pain. This process will be carried out three times in the same place and within an interval of 30 to 60 s, using the average of these three measurements.
Measurement of respiratory parameters through spirometry | immediately after the intervention/procedure/surgery
  First the subject is seated, the patient holds the spirometer horizontally in his right hand with the screen pointing upward. He puts the spirometer near his mouth and presses the operation button. You will hear a short beep. At the second beep, the subject takes in as much air as possible. Then place the mouthpiece of the spirometer in your mouth and blow as hard as you can for at least 1.5 seconds. The measurement will be repeated at least three times. One-minute intervals will be applied between these measurements to avoid fatigue of the respiratory muscles in the short term. We will measure the parameters of forced expiratory volume at one second (FEV1) and forced vital capacity (CVF).

OTHER OUTCOMES:
Schober test | 1 week after last intervention
  The Schober test measures the degree of elasticity of the spine, the coxofemoral joints or the hamstring muscles, taking into account that the overall mobility of the spine depends on all the segments that constitute it. It will be performed with the patient standing with his arms along the trunk. The therapist will stand on one side of the patient in a double feint facing towards him. With the help of a marker, the therapist makes a horizontal mark at the level of the S1 vertebra and another 10 cm above this first one. He asks the patient to lean forward and measures the distance between both marks. Next, he asks you again to extend the trunk and measures this distance again.
Fingers-Floor Distance (DDS) test | 1 week after last intervention
  This test is used to assess the elasticity of the spine. It will be performed with the patient standing with feet together and knees fully extended. The therapist will stand next to the patient in a squatting position to be able to make the resulting measurement with the help of a measuring tape. The therapist asks the patient to anteflexion the spine so that his arms, hands and fingers are fully extended and relaxed forward. In the same way, at the end of anteflexion the therapist must measure the distance between the tips of the fingers and the floor with a tape measure. If pain appears in the second part of the movement, one can think of the existence of a dysfunction of the lumbar spine or the sacroiliac joints. Likewise, if the symptoms are accentuated in the third part of anteflexion, the therapist may think of an alteration of the upper lumbar or thoracic spine.
Measurement of thoracic expansion | 1 week after last intervention
  It can be used as a method of evaluating the expansion of diaphragmatic breathing to quantify possible alterations in thoracic capacity and abdominal and chest wall compliance achieved by all expiratory and inspiratory muscles. By recording the expansion of the rib cage with a tape measure over the second intercostal space (axillary level), the xiphoid process, and the midpoint between the xiphoid process and the umbilicus (abdominal level), proficiency in diaphragmatic breathing can be demonstrated.It will be evaluated with cirtometry using a simple measuring tape, marked in centimeters, around the thorax and abdomen. With the patient standing and with their hands on their head, the patient will be asked to "inhale as much as possible" and "exhale as much as possible."
Pressure pain threshold (PPT) of the five lumbar vertebrae, quadratus lumborum and lumbar paravertebral | 1 week after last intervention
  using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer (quantitative v.), in the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L312. In the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L3. PPT measurements will be performed manually gradually until the patient begins to feel pain. This process will be carried out three times in the same place and within an interval of 30 to 60 s, using the average of these three measurements.
Measurement of respiratory parameters through spirometry | 1 week after last intervention
  First the subject is seated, the patient holds the spirometer horizontally in his right hand with the screen pointing upward. He puts the spirometer near his mouth and presses the operation button. You will hear a short beep. At the second beep, the subject takes in as much air as possible. Then place the mouthpiece of the spirometer in your mouth and blow as hard as you can for at least 1.5 seconds. The measurement will be repeated at least three times. One-minute intervals will be applied between these measurements to avoid fatigue of the respiratory muscles in the short term. We will measure the parameters of forced expiratory volume at one second (FEV1) and forced vital capacity (CVF).
Schober test | 4 weeks after last intervention
  The Schober test measures the degree of elasticity of the spine, the coxofemoral joints or the hamstring muscles, taking into account that the overall mobility of the spine depends on all the segments that constitute it. It will be performed with the patient standing with his arms along the trunk. The therapist will stand on one side of the patient in a double feint facing towards him. With the help of a marker, the therapist makes a horizontal mark at the level of the S1 vertebra and another 10 cm above this first one. He asks the patient to lean forward and measures the distance between both marks. Next, he asks you again to extend the trunk and measures this distance again.
Fingers-Floor Distance (DDS) test | 4 weeks after last intervention
  This test is used to assess the elasticity of the spine. It will be performed with the patient standing with feet together and knees fully extended. The therapist will stand next to the patient in a squatting position to be able to make the resulting measurement with the help of a measuring tape. The therapist asks the patient to anteflexion the spine so that his arms, hands and fingers are fully extended and relaxed forward. In the same way, at the end of anteflexion the therapist must measure the distance between the tips of the fingers and the floor with a tape measure. If pain appears in the second part of the movement, one can think of the existence of a dysfunction of the lumbar spine or the sacroiliac joints. Likewise, if the symptoms are accentuated in the third part of anteflexion, the therapist may think of an alteration of the upper lumbar or thoracic spine.
Measurement of thoracic expansion | 4 weeks after last intervention
  It can be used as a method of evaluating the expansion of diaphragmatic breathing to quantify possible alterations in thoracic capacity and abdominal and chest wall compliance achieved by all expiratory and inspiratory muscles. By recording the expansion of the rib cage with a tape measure over the second intercostal space (axillary level), the xiphoid process, and the midpoint between the xiphoid process and the umbilicus (abdominal level), proficiency in diaphragmatic breathing can be demonstrated.It will be evaluated with cirtometry using a simple measuring tape, marked in centimeters, around the thorax and abdomen. With the patient standing and with their hands on their head, the patient will be asked to "inhale as much as possible" and "exhale as much as possible."
Pressure pain threshold (PPT) of the five lumbar vertebrae, quadratus lumborum and lumbar paravertebral | 4 weeks after last intervention
  using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer (quantitative v.), in the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L312. In the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L3. PPT measurements will be performed manually gradually until the patient begins to feel pain. This process will be carried out three times in the same place and within an interval of 30 to 60 s, using the average of these three measurements.
Measurement of respiratory parameters through spirometry | 4 weeks after last intervention
  First the subject is seated, the patient holds the spirometer horizontally in his right hand with the screen pointing upward. He puts the spirometer near his mouth and presses the operation button. You will hear a short beep. At the second beep, the subject takes in as much air as possible. Then place the mouthpiece of the spirometer in your mouth and blow as hard as you can for at least 1.5 seconds. The measurement will be repeated at least three times. One-minute intervals will be applied between these measurements to avoid fatigue of the respiratory muscles in the short term. We will measure the parameters of forced expiratory volume at one second (FEV1) and forced vital capacity (CVF).
Schober test | 16 weeks after last intervention
  The Schober test measures the degree of elasticity of the spine, the coxofemoral joints or the hamstring muscles, taking into account that the overall mobility of the spine depends on all the segments that constitute it. It will be performed with the patient standing with his arms along the trunk. The therapist will stand on one side of the patient in a double feint facing towards him. With the help of a marker, the therapist makes a horizontal mark at the level of the S1 vertebra and another 10 cm above this first one. He asks the patient to lean forward and measures the distance between both marks. Next, he asks you again to extend the trunk and measures this distance again.
Fingers-Floor Distance (DDS) test | 16 weeks after last intervention
  This test is used to assess the elasticity of the spine. It will be performed with the patient standing with feet together and knees fully extended. The therapist will stand next to the patient in a squatting position to be able to make the resulting measurement with the help of a measuring tape. The therapist asks the patient to anteflexion the spine so that his arms, hands and fingers are fully extended and relaxed forward. In the same way, at the end of anteflexion the therapist must measure the distance between the tips of the fingers and the floor with a tape measure. If pain appears in the second part of the movement, one can think of the existence of a dysfunction of the lumbar spine or the sacroiliac joints. Likewise, if the symptoms are accentuated in the third part of anteflexion, the therapist may think of an alteration of the upper lumbar or thoracic spine.
Measurement of thoracic expansion | 16 weeks after last intervention
  It can be used as a method of evaluating the expansion of diaphragmatic breathing to quantify possible alterations in thoracic capacity and abdominal and chest wall compliance achieved by all expiratory and inspiratory muscles. By recording the expansion of the rib cage with a tape measure over the second intercostal space (axillary level), the xiphoid process, and the midpoint between the xiphoid process and the umbilicus (abdominal level), proficiency in diaphragmatic breathing can be demonstrated.It will be evaluated with cirtometry using a simple measuring tape, marked in centimeters, around the thorax and abdomen. With the patient standing and with their hands on their head, the patient will be asked to "inhale as much as possible" and "exhale as much as possible."
Pressure pain threshold (PPT) of the five lumbar vertebrae, quadratus lumborum and lumbar paravertebral | 16 weeks after last intervention
  using the Wagner Force TenTM Digital Force Gage model FPX 100 algometer (quantitative v.), in the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L312. In the center of the paravertebral spinal musculature bilaterally and perpendicular to the spinous process of L3. PPT measurements will be performed manually gradually until the patient begins to feel pain. This process will be carried out three times in the same place and within an interval of 30 to 60 s, using the average of these three measurements.
Measurement of respiratory parameters through spirometry | 16 weeks after last intervention
  First the subject is seated, the patient holds the spirometer horizontally in his right hand with the screen pointing upward. He puts the spirometer near his mouth and presses the operation button. You will hear a short beep. At the second beep, the subject takes in as much air as possible. Then place the mouthpiece of the spirometer in your mouth and blow as hard as you can for at least 1.5 seconds. The measurement will be repeated at least three times. One-minute intervals will be applied between these measurements to avoid fatigue of the respiratory muscles in the short term. We will measure the parameters of forced expiratory volume at one second (FEV1) and forced vital capacity (CVF).
Evaluation of quality of life using the SF-12 life questionnaire. (quantitative v.) | 16 weeks after last intervention
  The health-related quality of life questionnaire Short-Form 12-item (SF-12), which will be applied to determine the measure of health-related quality of life in the direct score and the optimal normalized values to evaluate the domains of physical and mental health. The evaluator will explain each of the items on the scales to the patient, and the patient will complete them in paper format in the presence of the evaluator to resolve any questions they may have. Later the evaluator will extract the scores. Scale of 12 questions in which each item of the scale evaluates different aspects on a scale from 0 (no quality of life) to 100 (highest quality of life). 100 being a result that indicates optimal health and 0 reflecting a state of very bad health.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Díaz-Mancha, PhD, Principal Investigator — University of Seville
Locations (1):
- Juan Antonio Díaz-Mancha, Seville, Seville, Spain

REFERENCES:
- [Derived] Vera-Serrano FJ, Vinolo-Gil MJ, Fernandez Seguin LM, Diaz-Mancha JA. Effects of diaphragmatic manual therapy on respiratory function in patients with non-specific low back pain: A randomized control trial. Respir Med. 2025 Nov;248:108394. doi: 10.1016/j.rmed.2025.108394. Epub 2025 Oct 4. PMID 41047009